CLINICAL TRIAL: NCT06140251
Title: Investigation of Biomarker Response to SGLT2 Inhibition Across Various Phenotypes of Heart Failure
Brief Title: Investigation of Biomarker Response to SGLT2 Inhibition in Heart Failure
Acronym: SiN-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Chris Watson, Dr, Queen's University, Belfast
Other Study IDs: 22063CW-UC
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac imaging; SGLT2; Biomarkers
MeSH Terms: conditions — Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be collected at both time points using a commercially available kit (SalivaBio Oral Swab Device, Salimetrics LLC, Carlsbad, CA, USA). Blood samples for novel biomarkers will be undergo centrifugation at 2500 g for 10 min with subsequent aliquoting and storage of plasma at -80 ∘C until required. Enzyme-linked immunosorbent assay (ELISA) based assays will be used to quantify levels of novel proteins as detailed below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sodium-glucose cotransporter 2 inhibitor — Patients identified with heart failure (both reduced ejection fraction and preserved) who are on optimal standard therapy and are candidates for treatment with SGLT2 inhibition will be identified from local heart failure databases, and local heart failure clinics. Following signed, informed consent and screening, patients will be allocated a first appointment where baseline clinical assessment and biomarker analysis will be obtained along with commencement on a SGLT2 inhibitor. Repeat assessment will be performed following a minimum period of 26 weeks.
  Other Names: SGLT2 inhibitors

SUMMARY:
This is a 26-week, open label, single-arm prospective evaluation of the effects of sodium glucose cotransporter 2 (SGLT2) inhibition on cardiac biomarkers, myocardial remodeling and patient reported outcomes in heart failure with both impaired and preserved left ventricular fraction.

DETAILED DESCRIPTION:
The primary aims of this study are to evaluate whether SGLT2 inhibition in patients with heart failure effects changes in novel cardiac biomarkers. This is an exploratory evaluation of novel cardiac pathways which may serve to establish, as of yet unknown, therapeutic mechanisms of action of SGLT2 inhibition in heart failure. Secondary aims include evaluation of changes in standard of care biomarkers following SGLT2 inhibition and changes in markers of cardiac remodeling as identified on echocardiography. Further exploratory analysis will seek to correlate changes in quantitative and qualitative heart failure outcomes with changes in both novel and standard of care cardiac biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent prior to any study specific procedures.
2. Male or female, between 40 and 90 years of age.
3. LVEF <50% on echocardiography or if >50%, co-existing structural markers of diastolic dysfunction must be present;

   * LA width (diameter) ≥3.8 cm or LA length ≥5.0 cm, or LA area ≥20 cm, or LA volume ≥55 mL or LA volume index ≥29 mL/m.
   * Left ventricular hypertrophy.
   * Markers of diastolic dysfunction as assessed by pulsed wave doppler echocardiography.
   * N-terminal pro-B-type natriuretic peptide (NT-proBNP) of at least 125pg per millilitre (or ≥365pg per millilitre if co-existing atrial fibrillation).
4. New York Heart Association (NYHA) class II, III, or IV symptoms.
5. On optimal tolerated evidence-based HF medications.
6. Patients may be ambulatory or recently hospitalized; however, must be >6 weeks post-discharge on stable diuretic therapy.

Exclusion Criteria:

1. Receiving therapy with an SGLT2 inhibitor > 6 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor.
2. Severe (eGFR <20 mL/min/1.73m2), unstable or rapidly progressing renal disease at the time of recruitment.
3. Type 1 diabetes mellitus
4. Recent hospitalisation < 1 month.
5. Symptomatic hypotension or systolic BP <95 mmHg at 2 out of 3 measurements
6. Symptomatic bradycardia or second or third-degree heart block without a pacemaker.
7. Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after recruitment.
8. Cardiomyopathy secondary to uncorrected primary valvular disease, infiltrative, arrhythmogenic or right ventricular dysplasia.
9. Significant comorbidity including; pulmonary lung disease requiring home oxygen or non-invasive ventilation, CTEPH or primary pulmonary hypertension.

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients identified with heart failure (both reduced ejection fraction and preserved) who are on optimal standard therapy and are candidates for treatment with SGLT2 inhibition will be identified from local heart failure databases, and local heart failure clinics. Following signed, informed consent and screening, patients will be enrolled into the trial.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether SGLT2 inhibition in heart failure produces changes in novel cardiac biomarkers. | 26 weeks
  Assessment of changes in levels of novel biomarkers associated with heart failure, cardiac remodeling, or response to SGLT2i, including; KIM-1, IGFBP7, TNFR, IL-6, collagen IV, MMP7, FN1, sST2, LRG1, Tetranectin, collagen XIV (Olink and ELISA based analysis). Additional novel biomarkers may be added to this investigatory panel as the trial continues.

SECONDARY OUTCOMES:
To evaluate if SGLT2 inhibition produces changes in markers of cardiac remodeling as assessed by echocardiography. | 26 weeks
  Changes in global longitudinal strain (GLS) (%) and left ventricular systolic function [LVEF (%)] as assessed on strain echocardiography.
To evaluate if SGLT2 inhibition produces changes in markers of cardiac remodeling as assessed by echocardiography. | 26 weeks
  Change in left ventricular end systolic volume index [LVESVi (mls/m2)], left ventricular end diastolic volume [LVEDVi (mls/m2)] and left atrial volume [LAVi (mls/m2)].
To evaluate if SGLT2 inhibition produces changes in markers of cardiac remodeling as assessed by diastolic parameters on echocardiography. | 26 weeks
  Change in left ventricular lateral e' (cm/s), septal e' (cm/s) and E/e' ratio obtained from echocardiography.
To evaluate changes in quantitative markers of heart failure outcomes following initiation of SGLT2 inhibition in heart failure. | 26 weeks
  Changes in standard care cardiac biomarkers following SGLT2 inhibition including, N-terminal prohormone of brain natriuretic peptide [NT-proBNP (ng/L)] and high sensitivity troponin [hs-TnT (ng/L)].
To evaluate changes in quantitative markers of heart failure outcomes following initiation of SGLT2 inhibition in heart failure. | 26 weeks
  Changes in standard care biomarker of inflammation following SGLT2 inhibition by measurement of serum C-reactive protein [CRP (mg/dL).
To evaluate changes in quantitative markers of heart failure outcomes following initiation of SGLT2 inhibition in heart failure. | 26 weeks
  Changes in standard care cardiac of diabetic biomarkers following SGLT2 inhibition using measurement of glycosylated haemoglobin [HbA1c (mmol/mol)].
To evaluate changes in quantitative markers of heart failure outcomes following initiation of SGLT2 inhibition in heart failure. | 26 weeks
  Changes in standard care biomarkers of cardiovascular risk following SGLT2 inhibition including lipid profile as assessed by serum cholesterol (mmol/L) and serum low density lipoprotein [LDL (mmol/L)].
To evaluate changes in qualitative markers of heart failure outcomes. | 26 weeks.
  Change in New York Heart Association (NYHA) score, classified on a scale I to IV, with a higher number indicating a worse outcome.
To evaluate changes in qualitative markers of heart failure outcomes. | 26 weeks.
  Change in Kansas-City Cardiomyopathy Questionnaire (KCCQ) score following initiation of SGLT2 inhibition in heart failure. It contains four subdomains: Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status. A change of 5 points on the scale scores, either as a group mean difference or an intra-individual change is defined as clinically significant.

OTHER OUTCOMES:
Exploratory evaluation of correlation of effect of SGLT2 inhibition on novel cardiac biomarkers with markers of cardiac remodeling. | 26 weeks.
  Correlation of log transformed delta change in novel cardiac biomarkers with global longitudinal strain [GLS (%)] and left ventricular ejection fraction [LVEF (%)].
Exploratory evaluation of correlation of effect of SGLT2 inhibition on novel cardiac biomarkers with markers of cardiac remodeling. | 26 weeks.
  Correlation of log transformed delta change in novel cardiac biomarkers with change in left ventricular end systolic volume index [LVESVi (mls/m2)], left ventricular end diastolic volume [LVEDVi (mls/m2)] and left atrial volume [LAVi (mls/m2)].
Exploratory evaluation of correlation of effect of SGLT2 inhibition on novel cardiac biomarkers with qualitive markers of heart failure outcomes. | 26 weeks.
  Correlation of log transformed delta change in novel cardiac biomarkers with change in Kansas-City Cardiomyopathy Questionnaire (KCCQ).
Exploratory evaluation of correlation of effect of SGLT2 inhibition on novel cardiac biomarkers with qualitive markers of heart failure outcomes. | 26 weeks.
  Correlation of log transformed delta change in novel cardiac biomarkers with change in Change in New York Heart Association (NYHA) score.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Watson, PHD, Study Chair — Queens University Belfast; Lana Dixon, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided